CLINICAL TRIAL: NCT03974516
Title: A Phase I Dose-Escalation Study in Healthy Volunteers to Evaluate the Safety and Tolerability Profiles of Careseng 1370
Brief Title: Careseng 1370 for Healthy Volunteers
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: This study was early terminated by the sponsor considering the difficulty of subject recruitment in the pandemic of COVID-19.
Sponsor: i Cure Biotech Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: Careseng 1370-01
Record Dates: First submitted 2019-05-30; First posted 2019-06-05 (Actual); Results first posted 2024-11-22 (Actual); Last update posted 2024-11-22 (Actual); Status verified 2024-09

CONDITIONS: Chemotherapy-induced Myelosuppression

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Careseng 1370 Level A (Experimental): Level A (1 sachet): 1 sachet before breakfast. Careseng 1370 granule 4,000 mg sachet consisted of 652 mg (16.3%, w/w) DS-1370 drug substance powder (dry extracts of Panax notoginseng stems and leaves)
  Interventions: Drug: Careseng 1370
- Careseng 1370 Level B (Experimental): Level B (2 sachets): 1 sachet before breakfast, 1 sachet before lunch. Careseng 1370 granule 4,000 mg sachet consisted of 652 mg (16.3%, w/w) DS-1370 drug substance powder (dry extracts of Panax notoginseng stems and leaves)
  Interventions: Drug: Careseng 1370
- Careseng 1370 Level C (Experimental): Level C (3 sachets): 1 sachet before breakfast, 2 sachets before lunch. Careseng 1370 granule 4,000 mg sachet consisted of 652 mg (16.3%, w/w) DS-1370 drug substance powder (dry extracts of Panax notoginseng stems and leaves)
  Interventions: Drug: Careseng 1370
- Careseng 1370 Level D (Experimental): Level D (1 sachet)(modified cohort): 1 sachet before breakfast on 1st, 3rd and 5th days.
  Careseng 1370 granule 4,000 mg sachet consisted of 652 mg (16.3%, w/w) DS-1370 drug substance powder (dry extracts of Panax notoginseng stems and leaves)
  Interventions: Drug: Careseng 1370

INTERVENTIONS:
Drug: Careseng 1370 — Careseng 1370 should be taken around 1 hour before meal.

SUMMARY:
This study will be performed in healthy volunteers in a conventional 3+3 dose-escalation design.

DETAILED DESCRIPTION:
Four cohorts (dose level A, B, C, and D) of up to 6 evaluable volunteers per cohort are planned to be sequentially accrued to receive Careseng 1370 1, 2, and 3 sachets per day, 4,000 mg/sachet before meal (starting from 1 sachet). At least 5 days of staggering and with the investigator's judgement of no safety concern will be required to administer the next volunteer for the first three volunteers of each cohort. The staggering time is counted from Day 1 of one volunteer to Day 1 of the next volunteer.

Careseng 1370 should be taken around 1 hour before meal. No volunteer is allowed to be assigned to more than 1 dose level. All dose escalation/de-escalation decisions will be made by the Data and Safety Monitoring Board (DSMB).

ELIGIBILITY:
Inclusion Criteria:

1. Adult aged between 20-40 years old (inclusive)
2. Physically and mentally healthy volunteer as confirmed by an interview, medical history, clinical examination, chest X-rays, and electrocardiogram. Volunteer with non-clinically significant signs or symptoms may be eligible at investigator's discretion.
3. Body Mass Index (BMI) between 18.5 and 24, inclusive (BMI will be calculated as weight in kilogram [kg]/(height in meters)2 [m2])
4. Clinically normal hematology, biochemistry and urinalysis determinations based on investigator's discretion. Volunteer with non-clinically significant signs or symptoms may be eligible at investigator's discretion.
5. Volunteer is willing and able to comply with study procedures and sign informed consent prior to initiation of any study-mandated procedures.

Exclusion Criteria:

1. Volunteer who has a history or evidence of a medical condition that would expose them to a risk of a significant adverse event or interfere with the assessments of safety or pharmacodynamics variables during the course of the trial, including but not limited to hepatic, renal, respiratory, cardiovascular, endocrine, immune, neurological, musculoskeletal or hematological disease as determined by the clinical judgment of the investigator
2. Volunteer has received any other investigational agent within 28 days prior to the first dose of study drug
3. Volunteer has taken or potentially takes any herbal medication/supplements/medicinal food, prescription medication and/or over-the-counter medication within 2 weeks prior to the first dose of study drug
4. Volunteer has alcohol, caffeine, grapefruit juice, or nicotine consumption within 24 hours prior to the first dose of study drug
5. Female volunteer of childbearing potential who:

   * is lactating; or
   * has positive pregnancy test result at eligibility checking; or
   * refuses to adopt at least two forms of birth control (at least one of which must be a barrier method) from Screening visit to Final visit.

   Note:

   Acceptable forms include:
   1. Established use of oral, injected or implanted hormonal methods of contraception.
   2. Placement of an intrauterine device (IUD) or intrauterine system (IUS).
   3. Barrier methods of contraception: Condom OR Occlusive cap (diaphragm or cervical/vault caps)
6. Male volunteer with female spouse/partners who are of childbearing potential refuses to adopt at least two forms of birth control (at least one of which must be a barrier method) from Screening visit until Final visit
7. Known or suspected allergy or hypersensitivity to any ingredients of study product
8. With history of stroke, myocardial infarction, or Coronary Artery Bypass Graft (CABG) surgery within the last 6 months prior to the screening visit
9. With history of cardiac failure (NYHA class 2 or above), unstable angina, or life-threatening arrhythmia within the last 6 months prior to the screening visit Note: NYHA = New York Heart Association
10. With blood pressures as systolic blood pressure < 90 mmHg or > 170 mmHg or diastolic blood pressure < 50 mmHg or > 120 mmHg at eligibility checking
11. History of psychiatric disorder
12. History of left ventricular outflow obstruction, such as aortic stenosis and hypertrophic cardiomyopathy
13. With a history of human immunodeficiency virus (HIV) infection or hepatitis B or C infection
14. Plan to receive surgery from Screening visit until Final visit
15. Known or suspected hypersensitivity to any component of Careseng 1370, including components in plants of genus Panax, Tween 80, Kolliphor® P188, Fujicalin, and ginseng flavor

Ages: 20 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 13 (Actual)
Dates: Start 2020-08-10 (Actual); Primary Completion 2022-03-11 (Actual); Study Completion 2022-03-11 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Taipei Medical University Hospital, Taipei, Taiwan

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: After the enrollment for Cohort A and Cohort B was completed, this study was early terminated by the sponsor considering the difficulty of subject recruitment in the pandemic of COVID-19. As a result, no subject was recruited to Cohort C and Cohort D.
Groups:
- Careseng 1370 Level A: Level A (1 sachet): 1 sachet before breakfast
  Careseng 1370: Careseng 1370 should be taken around 1 hour before meal.
  Careseng 1370 granule 4,000 mg sachet consisted of 652 mg (16.3%, w/w) DS-1370 drug substance powder (dry extracts of Panax notoginseng stems and leaves)
- Careseng 1370 Level B: Level B (2 sachets): 1 sachet before breakfast, 1 sachet before lunch.
  Careseng 1370: Careseng 1370 should be taken around 1 hour before meal.
  Careseng 1370 granule 4,000 mg sachet consisted of 652 mg (16.3%, w/w) DS-1370 drug substance powder (dry extracts of Panax notoginseng stems and leaves)
Period: Overall Study
Arm/Group | Careseng 1370 Level A | Careseng 1370 Level B
Started | 6 | 7 (There was one subject violating exclusion criteria 11 (history of psychiatric disorder) and was considered wrong entry.)
Completed | 6 | 7 (There was one subject violating exclusion criteria 11 (history of psychiatric disorder) and was considered wrong entry.)
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: After the enrollment for Cohort A and Cohort B was completed, this study was early terminated by the sponsor considering the difficulty of subject recruitment in the pandemic of COVID-19. As a result, no subject was recruited to Cohort C and Cohort D.
  There was one subject in Cohort B violating exclusion criteria 11 (history of psychiatric disorder) and was considered wrong entry.
Groups:
- Careseng 1370 Level A: Level A (1 sachet): 1 sachet before breakfast;
  Careseng 1370: Careseng 1370 should be taken around 1 hour before meal.
- Careseng 1370 Level B: Level B (2 sachets): 1 sachet before breakfast, 1 sachet before lunch
  Careseng 1370: Careseng 1370 should be taken around 1 hour before meal.
- Total: Total of all reporting groups
Arm/Group | Careseng 1370 Level A | Careseng 1370 Level B | Total
Number analyzed (Participants) | 6 | 7 | 13
Age, Continuous [Mean (Standard Deviation); unit: years] | 24.3 (2.25) | 26.0 (2.52) | 25.2 (2.45)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 2 | 6
  Male | 2 | 5 | 7
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 6 | 7 | 13
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 0 | 0 | 0
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  Taiwan | 6 | 7 | 13
Body Weight [Mean (Standard Deviation); unit: kg] | 62.3 (11.59) | 55.9 (8.31) | 58.9 (10.07)
Height [Mean (Standard Deviation); unit: cm] | 167.3 (9.81) | 162.4 (7.23) | 164.7 (8.52)
BMI [Mean (Standard Deviation); unit: kg/m^2] | 22.11 (1.572) | 20.90 (2.002) | 21.46 (1.851)

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Adverse Events (AEs) and/or Serious Adverse Events (SAEs)
Description: An AE is any untoward medical occurrence in a volunteer or clinical investigation participant administered a study medication and that does not necessarily have a causal relationship with this treatment. Laboratory abnormalities should not be recorded as AE unless determined to be clinically significant by Investigator.
  A SAE is defined as an AE meeting one of the following conditions:
  * Death during the period of protocol defined surveillance
  * Life Threatening Event (defined as a participant at immediate risk of death at the time of the event)
  * An event requiring in volunteer hospitalization or prolongation of existing hospitalization during the period of protocol defined surveillance
  * Results in congenital anomaly or birth defect
  * Results in a persistent or significant disability/incapacity
  * Based upon appropriate medical judgment, the event may jeopardize the participant and may require medical or surgical intervention to prevent one of the outcomes listed above.
Time Frame: Day -14 to Day 22
Population: Volunteers received any Careseng 1370
Measure: Count of Participants; unit: Participants
Arm/Group | Careseng 1370 Level A | Careseng 1370 Level B
Number analyzed (Participants) | 6 | 7
Participants
  Subjects with AE | 3 | 5
  Subjects with SAE | 0 | 0

2. Secondary Outcome: Number of Participants With no Change From Baseline to Applicable Post-dosing Visits in Body Weight (kg)
Description: *Baseline will be the value of measurement closest to and before start of IP administration.
  "Body weight unchanged from Baseline to Day X" indicates that the body weight on Day X minus the body weight at baseline has a 95% confidence interval that includes zero.
Time Frame: Day -14 to Day 22
Population: Volunteers received any Careseng 1370
  After the enrollment for Cohort A and Cohort B was completed, this study was early terminated by the sponsor considering the difficulty of subject recruitment in the pandemic of COVID-19. As a result, no subject was recruited to Cohort C and Cohort D.
  There was one subject violating exclusion criteria 11 (history of psychiatric disorder) and was considered wrong entry.
Measure: Count of Participants; unit: Participants
Arm/Group | Careseng 1370 Level A | Careseng 1370 Level B
Number analyzed (Participants) | 6 | 7
Participants
  Body weight unchanged from Baseline to Day 2 | 6 | 7
  Body weight unchanged from Baseline to Day 3 | 6 | 7
  Body weight unchanged from Baseline to Day 4 | 6 | 7
  Body weight unchanged from Baseline to Day 5 (Pre-dose) | 6 | 7
  Body weight unchanged from Baseline to Day 6 | 6 | 7
  Body weight unchanged from Baseline to Day 12 | 6 | 7
  Body weight unchanged from Baseline to Day 22 | 6 | 7

3. Secondary Outcome: Number of Participants With Clinical Laboratory Abnormalities
Description: The laboratory examinations include Hematology tests (CBC, PT and aPTT), Biochemistry (AST, ALP, ALT, bilirubin, creatinine, BUN, CRP, total protein, r-GT, lipid and electrolytes) and Urinalysis (pH, protein, RBC, WBC and urine cast).
  *Baseline will be the value of measurement closest to and before start of IP administration.
Time Frame: Day -14 to Day 22
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Careseng 1370 Level A | Careseng 1370 Level B
Number analyzed (Participants) | 6 | 7
Participants
  Lymphocytes (%) (Day 2), Clinically Significant Abnormalities | 0 | 1
  Lymphocytes (%) (Day 12), Clinically Significant Abnormalities | 1 | 0
  Lymphocyte Count (10^9/L) (Day 2), Clinically Significant Abnormalities | 0 | 1
  Lymphocyte Count (10^9/L) (Day 12), Clinically Significant Abnormalities | 1 | 0
  International normalized ratio (Day5, 4 hours post dosing), Clinically Significant Abnormalities | 1 | 0
  APTT (Day 1, 8 hours post dosing), Clinically Significant Abnormalities | 1 | 0
  APTT (Day 2), Clinically Significant Abnormalities | 1 | 0
  APTT (Day 3), Clinically Significant Abnormalities | 1 | 0
  APTT (Day 4), Clinically Significant Abnormalities | 1 | 0
  APTT (Day 5, Pre-dose), Clinically Significant Abnormalities | 1 | 0
  APTT (Day 5, 4 hours post dosing), Clinically Significant Abnormalities | 1 | 0
  APTT (Day 6), Clinically Significant Abnormalities | 1 | 0
  APTT (Day 22), Clinically Significant Abnormalities | 1 | 0
  Lipase (U/L) (Day 1, 8 hours post dosing), Clinically Significant Abnormalities | 0 | 1
  Lipase (U/L) (Day 3), Clinically Significant Abnormalities | 0 | 1
  Lipase (U/L) (Day 6), Clinically Significant Abnormalities | 0 | 2
  Lipase (U/L) (Day 22), Clinically Significant Abnormalities | 0 | 1

4. Secondary Outcome: Number of Participants With Vital Signs Abnormalities
Description: Vital signs measurement will consist of systolic/diastolic blood pressure, respiratory rate, pulse rate or heart rate, and body temperature.
Time Frame: Day -14 to Day 22
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Groups:
- Careseng 1370 Level A: Level A (1 sachet): 1 sachet before breakfast
  Careseng 1370: Careseng 1370 should be taken around 1 hour before meal.
Arm/Group | Careseng 1370 Level A | Careseng 1370 Level B
Number analyzed (Participants) | 6 | 7
Participants | 0 | 0

5. Secondary Outcome: Number of Participants With Physical Examination Abnormalities
Description: Physical examination will include the following items: general appearance, skin, eyes, ears, nose, throat, head and neck, heart, chest and lungs, abdomen, extremities, lymph nodes, musculoskeletal, neurological and others.
Time Frame: Day -14 to Day 22
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Careseng 1370 Level A | Careseng 1370 Level B
Number analyzed (Participants) | 6 | 7
Participants
  Extremities (Day 12) | 0 | 1
  Skin (Day 22) | 0 | 1

6. Secondary Outcome: Plasma Concentration of Marker Ingredients in Careseng 1370, 20(S)-Protopanaxadiol (PPD) and Its Metabolites
Description: Maximum plasma concentration (Cmax) of PPD and its metabolites, M-C1, and M-C2.
Time Frame: Day 2 to Day 8
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Careseng 1370 Level A | Careseng 1370 Level B
Number analyzed (Participants) | 6 | 7
ng/mL
  PPD at Day 2 pre-dose | 11.2 (3.34) | 42.9 (6.15)
  PPD at Day 3 pre-dose | 11.3 (5.70) | 75.8 (33.6)
  PPD at Day 4 pre-dose | 19.8 (13.3) | 63.0 (41.0)
  PPD at Day 5 pre-dose | 22.2 (22.3) | 57.1 (42.4)
  PPD at Day 5 0.5 hr post-dose | 65.8 (31.6) | 121 (68.7)
  PPD at Day 5 1 hr post-dose | 71.5 (35.8) | 146 (78.4)
  PPD at Day 5 2 hr post-dose | 148 (73.0) | 248 (94.0)
  PPD at Day 5 4 hr post-dose: number analyzed (Participants) | 6 | 6
  PPD at Day 5 4 hr post-dose | 130 (129) | 205 (116)
  PPD at Day 5 4.5 hr post-dose: number analyzed (Participants) | 0 | 7
  PPD at Day 5 4.5 hr post-dose |  | 209 (120)
  PPD at Day 5 5 hr post-dose: number analyzed (Participants) | 0 | 7
  PPD at Day 5 5 hr post-dose |  | 257 (117)
  PPD at Day 5 6 hr post-dose | 83.2 (70.8) | 488 (149)
  PPD at Day 5 7 hr post-dose: number analyzed (Participants) | 0 | 7
  PPD at Day 5 7 hr post-dose |  | 485 (224)
  PPD at Day 5 8 hr post-dose: number analyzed (Participants) | 0 | 7
  PPD at Day 5 8 hr post-dose |  | 365 (241)
  PPD at Day 5 9 hr post-dose: number analyzed (Participants) | 0 | 7
  PPD at Day 5 9 hr post-dose |  | 319 (222)
  PPD at Day 5 10 hr post-dose: number analyzed (Participants) | 0 | 7
  PPD at Day 5 10 hr post-dose |  | 253 (186)
  PPD at Day 5 12 hr post-dose | 34.2 (19.3) | 184 (137)
  PPD at Day 5 16 hr post-dose: number analyzed (Participants) | 0 | 7
  PPD at Day 5 16 hr post-dose |  | 107 (74.4)
  PPD at Day 6 | 20.6 (11.3) | 71.1 (40.7)
  PPD at Day 7 | 10.4 (5.09) | 32.0 (19.1)
  PPD at Day 8 | 6.37 (4.25) | 17.5 (10.3)
  M-C1 at Day 2 pre-dose | 29.1 (14.5) | 173 (85.6)
  M-C1 at Day 3 pre-dose | 35.9 (18.2) | 301 (275)
  M-C1 at Day 4 pre-dose | 64.5 (37.5) | 187 (192)
  M-C1 at Day 5 pre-dose | 46.9 (34.6) | 215 (285)
  M-C1 at Day 5 0.5 hr post-dose | 149 (41.2) | 296 (274)
  M-C1 at Day 5 1 hr post-dose | 187 (48.1) | 390 (334)
  M-C1 at Day 5 2 hr post-dose | 358 (97.5) | 570 (308)
  M-C1 at Day 5 4 hr post-dose | 351 (180) | 670 (484)
  M-C1 at Day 5 4.5 hr post-dose: number analyzed (Participants) | 0 | 7
  M-C1 at Day 5 4.5 hr post-dose |  | 638 (492)
  M-C1 at Day 5 5 hr post-dose: number analyzed (Participants) | 0 | 7
  M-C1 at Day 5 5 hr post-dose |  | 671 (497)
  M-C1 at Day 5 6 hr post-dose | 260 (131) | 926 (394)
  M-C1 at Day 5 7 hr post-dose: number analyzed (Participants) | 0 | 7
  M-C1 at Day 5 7 hr post-dose |  | 1040 (411)
  M-C1 at Day 5 8 hr post-dose: number analyzed (Participants) | 0 | 7
  M-C1 at Day 5 8 hr post-dose |  | 934 (487)
  M-C1 at Day 5 9 hr post-dose: number analyzed (Participants) | 0 | 7
  M-C1 at Day 5 9 hr post-dose |  | 925 (567)
  M-C1 at Day 5 10 hr post-dose: number analyzed (Participants) | 0 | 7
  M-C1 at Day 5 10 hr post-dose |  | 816 (515)
  M-C1 at Day 5 12 hr post-dose | 139 (69.4) | 673 (508)
  M-C1 at Day 5 16 hr post-dose: number analyzed (Participants) | 0 | 7
  M-C1 at Day 5 16 hr post-dose |  | 411 (372)
  M-C1 at Day 6 | 51.9 (17.2) | 247 (295)
  M-C1 at Day 7 | 12.8 (4.44) | 59.3 (86.8)
  M-C1 at Day 8 | 3.58 (2.46) | 14.1 (18.7)
  M-C2 at Day 2 pre-dose | 1.16 (0.598) | 5.33 (2.21)
  M-C2 at Day 3 pre-dose | 1.01 (0.785) | 12.2 (12.8)
  M-C2 at Day 4 pre-dose | 2.01 (0.883) | 7.44 (6.87)
  M-C2 at Day 5 pre-dose | 2.55 (3.47) | 6.07 (6.06)
  M-C2 at Day 5 0.5 hr post-dose | 14.9 (6.08) | 17.4 (10.4)
  M-C2 at Day 5 1 hr post-dose | 21.6 (8.92) | 30.8 (15.4)
  M-C2 at Day 5 2 hr post-dose | 43.4 (19.0) | 52.6 (12.3)
  M-C2 at Day 5 4 hr post-dose: number analyzed (Participants) | 6 | 6
  M-C2 at Day 5 4 hr post-dose | 40.9 (30.4) | 55.7 (27.6)
  M-C2 at Day 5 4.5 hr post-dose: number analyzed (Participants) | 0 | 7
  M-C2 at Day 5 4.5 hr post-dose |  | 52.5 (32.9)
  M-C2 at Day 5 5 hr post-dose: number analyzed (Participants) | 0 | 7
  M-C2 at Day 5 5 hr post-dose |  | 57.4 (32.2)
  M-C2 at Day 5 6 hr post-dose | 26.7 (20.4) | 89.8 (25.4)
  M-C2 at Day 5 7 hr post-dose: number analyzed (Participants) | 0 | 7
  M-C2 at Day 5 7 hr post-dose |  | 105 (34.2)
  M-C2 at Day 5 8 hr post-dose: number analyzed (Participants) | 0 | 7
  M-C2 at Day 5 8 hr post-dose |  | 87.1 (38.0)
  M-C2 at Day 5 9 hr post-dose: number analyzed (Participants) | 0 | 7
  M-C2 at Day 5 9 hr post-dose |  | 75.3 (38.3)
  M-C2 at Day 5 10 hr post-dose: number analyzed (Participants) | 0 | 7
  M-C2 at Day 5 10 hr post-dose |  | 60.4 (34.6)
  M-C2 at Day 5 12 hr post-dose | 6.24 (3.72) | 38.7 (27.7)
  M-C2 at Day 5 16 hr post-dose: number analyzed (Participants) | 0 | 7
  M-C2 at Day 5 16 hr post-dose |  | 16.8 (14.9)
  M-C2 at Day 6 | 2.29 (1.05) | 7.14 (6.51)
  M-C2 at Day 7 | 0.188 (0.459) | 1.86 (2.10)
  M-C2 at Day 8 | 0 (0) | 0.325 (0.861)

7. Secondary Outcome: Participants With Abnormal Sinus Rhythm
Description: Sinus rhythm was measured by 12-lead EKG
Time Frame: Day -14 to Day 22
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Groups:
- Careseng 1370 Level B: Level B (2 sachets): 1 sachet before breakfast, 1 sachet before lunch.
  Careseng 1370: Careseng 1370 should be taken around 1 hour before meal.
Arm/Group | Careseng 1370 Level A | Careseng 1370 Level B
Number analyzed (Participants) | 6 | 7
Participants
  Baseline | 6 | 0
  Day 1, 1 hour post dosing | 3 | 0
  Day 1, 4 hour post dosing | 3 | 0
  Day 1, 8 hour post dosing | 1 | 0
  Day 1, 12 hour post dosing | 1 | 0
  Day 2, pre-dose | 2 | 0
  Day 2, 1 hour post dosing | 1 | 0
  Day 3, pre-dose | 2 | 0
  Day 3, 1 hour post dosing | 2 | 0
  Day 4, pre-dose | 1 | 0
  Day 4, 1 hour post dosing | 1 | 0
  Day 5, pre-dose | 4 | 0
  Day 5, 1 hour post dosing | 4 | 0
  Day 5, 4 hours post dosing | 2 | 0
  Day 5, 8 hours post dosing | 1 | 0
  Day 5, 12 hours post dosing | 1 | 0
  Day 6 | 0 | 0
  Day 12 | 0 | 0
  Day 22 | 2 | 0

8. Secondary Outcome: Significantly Abnormal Ventricular Rate Compared to Baseline
Description: Ventricular rate was measured by EKG.
Time Frame: Day -14 to Day 22
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: beats/min
Arm/Group | Careseng 1370 Level A | Careseng 1370 Level B
Number analyzed (Participants) | 6 | 7
beats/min
  Day 1, 4 hours post dosing - Baseline | 6.50 (12.755) | 9.29 (9.861)
  Day 5, 1 hour post dosing - Baseline | -1.00 (4.382) | 7.57 (5.350)
  Day 5, 4 hours post dosing - Baseline | 6.33 (6.022) | 4.57 (10.581)
  Day 5, 8 hours post dosing - Baseline | 10.00 (8.367) | 6.00 (9.147)
  Day 5, 12 hours post dosing - Baseline | 10.67 (8.091) | 5.86 (11.276)
  Day 12 - Baseline | 11.50 (9.375) | 10.29 (7.952)

9. Secondary Outcome: Significantly Abnormal PR, QRS, QT, QTc Intervals Compared to Baseline
Description: PR, QRS, QT and QTc intervals were measured by EKG.
Time Frame: Day -14 to Day 22
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: msec
Arm/Group | Careseng 1370 Level A | Careseng 1370 Level B
Number analyzed (Participants) | 6 | 7
msec
  PR Interval (msec) (Day 1, 4 hours post dosing - Baseline) | 0.00 (10.863) | -16.57 (25.045)
  PR Interval (msec) (Day 1, 12 hours post dosing - Baseline) | -5.17 (3.430) | -10.00 (19.545)
  PR Interval (msec) (Day 2, Pre-dose - Baseline) | -2.00 (7.403) | -12.57 (3.823)
  PR Interval (msec) (Day 5, Pre-dose - Baseline) | 3.67 (6.623) | -16.57 (14.547)
  PR Interval (msec) (Day 5, 4 hours post dosing - Baseline) | 2.67 (7.090) | -16.14 (13.582)
  QRS Interval (msec) (Day 12 - Baseline) | -2.17 (5.037) | -4.29 (3.684)
  QT Interval (msec) (Day 1, 8 hours post dosing - Baseline) | -21 (23.673) | -9.71 (23.655)
  QT Interval (msec) (Day 5, 12 hours post dosing - Baseline) | -25.67 (13.171) | -7.86 (40.544)
  QT Interval (msec) (Day 12 - Baseline) | -23.50 (18.229) | -17.43 (25.999)
  QTc Interval (msec) (Day 1, 4 hours post dosing - Baseline) | 1.83 (12.576) | 16.71 (13.937)
  QTc Interval (msec) (Day 1, 12 hours post dosing - Baseline) | 7.83 (5.947) | 16.57 (28.213)
  QTc Interval (msec) (Day 3, Pre-dose - Baseline) | 6.00 (13.914) | 15.57 (13.563)
  QTc Interval (msec) (Day 4, Pre-dose - Baseline) | 13.33 (11.759) | 7.29 (19.440)
  QTc Interval (msec) (Day 6 - Baseline) | 8.50 (14.923) | 8.71 (8.693)

10. Other Pre Specified Outcome: Number of Participants With Abnormal Immune Profile
Description: Immune profile includes percentages of CD3+, CD3+/CD4+, CD3+/CD8+, CD19+, CD16+/CD56+, and CD4/CD8 ratio
Time Frame: Day -14 to Day 22
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Careseng 1370 Level A | Careseng 1370 Level B
Number analyzed (Participants) | 6 | 7
Participants
  CD3+ (%) | 0 | 0
  CD3+/CD4+ (%) | 0 | 0
  CD3+/CD8+ (%) | 0 | 0
  CD19+ (%) | 0 | 0
  D16+/CD56+ (%) | 0 | 0
  CD4/CD8 Ratio | 0 | 0

ADVERSE EVENTS:
Time Frame: Day -14 to Day 22
Arm/Group | Careseng 1370 Level A | Careseng 1370 Level B
All-Cause Mortality (participants affected / at risk) | 0/6 | 0/7
Serious Adverse Events (participants affected / at risk) | 0/6 | 0/7
Other Adverse Events (participants affected / at risk) | 3/6 | 5/7
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Careseng 1370 Level A (N=6) | Careseng 1370 Level B (N=7)
Lipase increased (Investigations) | 0 (0) | 3 (5)
Activated partial thromboplastin time prolonged (Investigations) | 2 (3) | 0 (0)
Lymphocyte count decreased (Investigations) | 1 (1) | 1 (1)
Prothrombin time prolonged (Investigations) | 1 (1) | 0 (0)
Abdominal distension (Gastrointestinal disorders) | 0 (0) | 1 (1)
Dermatitis allergic (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)

LIMITATIONS AND CAVEATS:
Early termination leading to small numbers of subjects analyzed; wrong entry of one subject in dose level B leading to a skewed population.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less

DOCUMENTS (2):
  • Study Protocol (2020-09-18): https://cdn.clinicaltrials.gov/large-docs/16/NCT03974516/Prot_000.pdf
  • Statistical Analysis Plan (2022-09-08): https://cdn.clinicaltrials.gov/large-docs/16/NCT03974516/SAP_001.pdf